CLINICAL TRIAL: NCT04272749
Title: Determining Perceptions of 'Milk': Investigating Consumer Understanding of Dairy Milk and Plant-based Milk Alternatives
Brief Title: Consumer Perceptions of Milk Beverages
Acronym: CMK2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinical Nutrition Research Center, Illinois Institute of Technology (Industry)
Collaborators: Food and Drug Administration (FDA) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2019-059
Record Dates: First submitted 2020-02-13; First posted 2020-02-17 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: Consumer Behavior
Keywords: milk; dairy; plant-based milk alternatives; consumer choices; consumer behavior
MeSH Terms: conditions — Consumer Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dairy and non-dairy milks (Experimental): Questionnaires and consumption behaviors of dairy and non-dairy milks
  Interventions: Behavioral: Assess opinons on the milk beverages

INTERVENTIONS:
Behavioral: Assess opinons on the milk beverages — Questionnaires and consumption behaviors of dairy and non-dairy milks, including whole, 2% fat, 1% fat, skim, unsweetened almond, sweetened almond, unsweetened coconut, sweetened coconut, unsweetened soy, sweetened soy, unsweetened rice, and sweetened rice.....

SUMMARY:
The objectives of this study are to:

1. Investigate and describe perceptions of nutrient content, including calories, of plant-based milks and dairy milks without food labels (ie., no Ingredient or Nutrition Facts label) and how this impacts consumption choice.
2. Determine understanding of nutrient content, including calories, of plant-based milks and dairy milks after given access to food labels (ie., Ingredient or Nutrition Facts label) and how this impacts consumption choice.
3. Assess influence of age, gender, economic status, and race/ethnicity on results.

DETAILED DESCRIPTION:
The proposed study is to evaluate the nutrient content understanding of subjects before and after exposure to nutrition facts and ingredients list labels, along with the decision-making behind consumption choices. Before the activity, subjects will complete a consumer choice questionnaire and an eating habits questionnaire, which evaluates grocery shopping patterns and typical 'milk' beverage preferences of subjects prior to participation in the activity.

Subjects will be presented with several 'milk' products in a four-section activity. Carton set-up will vary between sections in terms of number and order. The order the cartons will be set up on the tables will be randomized for each subject in order to avoid having results attributed to the order the cartons are seen. In order to make a smooth randomization process, each carton with has a number sticker on it, such as '#1' '#2' and so on. If carton '#1' is almond milk in section I, it will remain carton '#1' for all subjects during section I - only the order that the cartons are placed will change. Each of the four sections of the activity will take place in its own cubicle. Subjects will be able to look at, move around, and compare cartons while answering questions for that section's respective questionnaire booklet. There will be no time limit on questionnaires. Questions in the booklet will be separated onto different pages in order to prevent subjects from looking back at previous answers and/or changing answers due to surrounding questions. Questionnaires throughout the four sections will assess consumer perceptions of nutrient content of 'milk' beverages before and after exposure to nutrition labels, exposure to varieties of 'milk,' and an ingestion component - the requirement to choose one smoothie in front of a 'milk' carton to consume. All cartons will remain unbranded throughout the activity. The difference between labeled and unlabeled cartons will be only the presence or absence, respectively, of a nutrition facts table and ingredients list on the side of the carton.

II. Study Subjects Subjects will be recruited through online advertisements, flyers distributed throughout the university and local communities, and word of mouth. Interested individuals can either click a link or scan a QR code to a secure online pre-screen survey available in online advertisements and on flyers, or will be directed to the secure online pre-screen survey by phone and/or email through using the contact information provided to the subject on the online advertisements and flyers. Based upon this initial screening outcome, subjects will be contacted to schedule their study visit. Upon arrival to the study visit, subjects will have their birth date and hunger level confirmed by study personnel. Hunger level will be analyzed through a Visual Analogue Scale (VAS) question. Subjects that mark a vertical line on the VAS that is under 25mm or over 75mm, meaning extreme fullness or extreme hunger, respectively, will be dismissed from the lab and are able to return at another time. One hundred (n=100) subjects will be recruited.

III. Study Procedures Recruited subjects must meet all eligibility criteria (age requirement, no allergies that could produce bias in choice during this study); sign and date a written Institutional Review Board (IRB) approved Informed Consent Form prior to any study procedures, and be willing and able to comply with study schedule and procedures. Subjects will also be asked to fast for two (2) hours before coming to our site - this means no eating or drinking other than water. During the screening visit, which includes confirming age and collecting basic health information (weight, height, body composition), participants will also complete questionnaires relating to eating habits and choice patterns in purchasing, including general questions about dairy milks and plant-based milk alternatives to assess consumption preferences. These will not be used for exclusion, but rather to characterize population included in the study from a general health standpoint. These answers will allow for understanding of selection bias when comparing those who do and do not complete the study. Subjects will be required to drink a smoothie containing strawberries and banana during their visit at the CNRC.

IV. Study Visit After completion of the initial online pre-screen questionnaire, eligible subjects will be provided the option to schedule a study visit time, meaning a time to come into the CNRC to complete the study.

The activity portion will be divided into four sections. Throughout this study, font, font size, and color will be standardized among all cartons. In the first section, the participant will be presented with five brand-less, unlabeled cartons: each of the five cartons will have only one of either a cow, almond, soy, rice, and coconut sticker on them, along with a number given to each carton for randomization purposes. In this section, the varieties in plant-based milk alternatives (sweetened and unsweetened) and the varieties in dairy milks (whole, 2%, 1%, and skim) will not be shown. A questionnaire booklet will be given to subjects, which will ask about word associations (the first words or phrases that come to mind when thinking of each type of 'milk' beverage) and preferences. This section serves to assess opinions on the beverages in the absence of variety and nutrition labeling. The second section introduces variety in that 12 brand-less, unlabeled cartons will have only a name and number sticker on them: whole, 2% fat, 1% fat, skim, unsweetened almond, sweetened almond, unsweetened coconut, sweetened coconut, unsweetened soy, sweetened soy, unsweetened rice, and sweetened rice will be shown. A questionnaire will be given to subjects, which will ask about preferences and nutrient content associations, along with interfering questions that are still of interest in order to avoid asking the nutrient association questions immediately after one another. The third and fourth sections will have the same 12 brand-less cartons, except all cartons will now have a nutrition facts and ingredients list label on their side. A questionnaire booklet will ask about preferences and potential standout information to the subject after the viewing of the nutrition labels. In the fourth section, the questionnaire booklet will ask about preferences and see if the decision-making process to consume a 'milk' beverage differs from that of only hypothetically choosing a 'milk' beverage. There will be a strawberry banana smoothie in a cup in front of each of the 'milk' cartons and subjects will answer the section's questionnaire before consuming the smoothie of their choice. Only the fourth section of the activity will require consumption of a 'milk' beverage; sections one, two, and three will not involve any smoothie consumption. Subjects will consume 2 ounces (oz) of the beverage they choose. These beverages will all be made of the same recipe containing strawberries, bananas, and water in the metabolic kitchen using appropriate standard food safety protocols. Each of the various 'milk' cartons will have a smoothie placed in front of it so that the subject chooses the smoothie they associate with that particular 'milk' carton. The second section will assess consumer opinions in the presence of variety without exposure to nutrition labeling, the third section will assess those opinions after exposure to nutrition labeling, and the fourth section will assess if those opinions differ when ingestion is added into the activity. Each subject will go through sections 1-4 in the same order. Upon completion of the activity, subjects will complete a post-screen to re-assess nutrient associations and opinions on dairy milk and plant-based milk alternatives after the activity compared to before the activity.

ELIGIBILITY:
Inclusion Criteria

* Able to provide informed consent and comply with study procedures

Exclusion Criteria

* Under 18 years old
* Lactose, cow's milk protein, and/or dairy intolerance
* Cow's milk protein and/or dairy allergy
* Nut allergy
* Vegan or vegetarian that excludes dairy products
* Strawberry and/or banana allergy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2019-12-16 (Actual); Primary Completion 2020-11-24 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Opinions on the beverages in the absence of variety and nutrition labeling via questionnaire | 3 minutes
  the participant will be presented with five brandless, unlabeled cartons: each of the five cartons will have only one of either a cow, almond, soy, rice, and coconut sticker on them. A questionnaire booklet will be given to subjects at the end of the three-minute timer including questions about word associations (the first words that come to mind when thinking of each type of 'milk' beverage) and preferences.
Preferences and potential standout information to the subject after the viewing of the nutrition labels via questionnaire | 20 minutes
  12 brandless, unlabeled cartons will have only a name and number sticker on them: whole, 2% fat, 1% fat, skim, unsweetened almond, sweetened almond, unsweetened coconut, sweetened coconut, unsweetened soy, sweetened soy, unsweetened rice, and sweetened rice will be shown, with and without nutrition facts and ingredients list label on their side.
Preferences for consumption via behavior assessment | 3 minutes
  There will be a strawberry banana smoothie in a cup in front of each of the 'milk' cartons and subjects will have the three-minute timer to further assess cartons before choosing which of the beverages is their pick to consume.

CONTACTS AND LOCATIONS:
Overall Officials: Britt M Burton-Freeman, Ph.D, Principal Investigator — Illinois Insititute of Technology
Locations (1):
- Clinical Nutrition Research Center, Chicago, Illinois, United States